CLINICAL TRIAL: NCT04710368
Title: Effect of Evolocumab on Coronary Plaque Characteristics: a Multimodality Imaging Study
Brief Title: Effect of Evolocumab on Coronary Plaque Characteristics
Acronym: YELLOW III
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Annapoorna Kini (Other)
Responsible Party: Sponsor-Investigator, Annapoorna Kini, Professor of Medicine, Cardiology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 20-2935
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Coronary Plaque; Optical Coherence Tomography; Near-Infrared Spectroscopy; Evolocumab; Statin
MeSH Terms: conditions — Coronary Artery Disease | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: The study team will screen patients scheduled for elective PCI, who are receiving statin therapy for at least 4 weeks with acceptable LDL-C levels. Patients with non-obstructive lesion (30-50% stenosis) by angiography and lipid-rich plaque with lipid arc >90° and minimal fibrous cap thickness ≤ 120 µm detected by OCT will comprise the final study population. Serial NIRS/IVUS and OCT imaging will be performed in a non-target lesions, first during PCI and subsequently after 26 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Evolocumab subcutaneously administered 140 mg every 2 weeks for 26 weeks
  Interventions: Drug: Evolocumab Injections

INTERVENTIONS:
Drug: Evolocumab Injections — Administered on day 1 (the day of the first treatment) and through week 26 with a personal injector or prefilled auto injector/pens.
  Other Names: Repatha

SUMMARY:
The aim of the study is to assess the effect of evolocumab on coronary plaque morphology using intravascular imaging and gene expression analysis of peripheral blood mononuclear cells (PBMC) in patients with stable CAD on maximally tolerated statin therapy. The study combines multi-modality intravascular imaging approaches and transcriptomic based machine learning algorithms to uncover molecular mechanisms responsible for the beneficial changes in atherosclerotic lesions of patients treated with evolocumab. The primary end-points are the changes from baseline to follow-up in (1) the minimal fibrous cap thickness (FCT) assessed by optical coherence tomography (OCT) and (2) maxLCBI4mm assessed by near-infrared spectroscopy (NIRS) after 26 weeks of evolocumab. The secondary endpoints are the changes in (1) the maximal lipid arc, lipid length, lipid volume index, macrophage accumulation and calcification by OCT; (2) PAV and TAV defined by intravascular ultrasound (IVUS) and (3) Changes in PBMC gene expression.

DETAILED DESCRIPTION:
The single center single arm study will be performed in the Cardiac Catheterization laboratory of the Mount Sinai Hospital, New York, NY. After informed consent, patients undergoing clinically indicated elective PCI with a non-obstructive lesion and optimal background statin therapy will be eligible screening. Non-obstructive lesions (30-50% stenosis) identified by angiography in a non-culprit vessel with lipid-rich plaque will be studied. Subjects will receive evolocumab (Repatha) 140 mg subcutaneously every 2 weeks for 26 weeks. Serial NIRS/IVUS and OCT imaging will be performed in the non-obstructive lesions, first during PCI and subsequently after 26 weeks. A total of 25ml of blood will be drawn from the sheath during angiography for transcriptomic profiling of PBMC.

ELIGIBILITY:
Inclusion criteria:

* Men or women aged 18 years or older at screening who signed written Informed Consent
* Patients with coronary artery disease undergoing cardiac catheterization and PCI for a target lesion and also have a non-obstructive lesion (30-50% stenosis) identified by angiography
* Patients who are not candidates for PCI or CABG currently or over the next 12 months, in the opinion of the investigator
* Patients treated with statins for at least 4 weeks with LDL-C level ≥ 80 mg/dL for low- or moderate -intensity statin use and ≥ 60 mg/dL for high-dose statin. Patients with history of statin intolerance and LDL-C ≥ 100 mg/dL.
* Angiographic criteria: 30-50% reduction of lumen diameter in addition to the target lesion accessible by the OCT catheter. The target segment should not have a history of percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG), and may not be a bypass graft.
* OCT criteria: target segment should have a lipid-rich plaque with lipid arc >90° and fibrous cap thickness ≤120 µm.
* Women of childbearing potential must agree to be on an acceptable method of birth control/contraceptive

Exclusion criteria:

* Patients who have acute myocardial infarction (Q wave or non-Q wave with CK-MB > 5 times above the upper normal (31.5 ng/ml) within 72 hours)
* Patients who are in cardiogenic shock
* Patients with left main disease, in-stent restenotic lesions or patients requiring coronary artery bypass graft surgery
* Patients with elevated CK-MB (>6.3 ng/ml) or Tnl (>0.5 ng/ml)
* Patients with platelet count < 100,000 cell/mm3
* Patients who have co-morbidity which reduces life expectancy to one year
* Patients who are currently participating in another investigational drug/device study
* Patients with liver disease
* Patient with creatinine > 2.0 mg/dL
* Pregnant women and women of childbearing potential who intend to have children during the duration of the trial
* Patients having undergone heart transplantation, or those that may undergo heart transplantation during the study period
* Patients with active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nissen SE, Stroes E, Dent-Acosta RE, Rosenson RS, Lehman SJ, Sattar N, Preiss D, Bruckert E, Ceska R, Lepor N, Ballantyne CM, Gouni-Berthold I, Elliott M, Brennan DM, Wasserman SM, Somaratne R, Scott R, Stein EA; GAUSS-3 Investigators. Efficacy and Tolerability of Evolocumab vs Ezetimibe in Patients With Muscle-Related Statin Intolerance: The GAUSS-3 Randomized Clinical Trial. JAMA. 2016 Apr 19;315(15):1580-90. doi: 10.1001/jama.2016.3608. PMID 27039291
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Connolly CK. Lung function testing. Respir Med. 1994 Nov;88(10):795-6. doi: 10.1016/s0954-6111(05)80207-0. No abstract available. PMID 7846344
- [Background] Kini AS, Vengrenyuk Y, Shameer K, Maehara A, Purushothaman M, Yoshimura T, Matsumura M, Aquino M, Haider N, Johnson KW, Readhead B, Kidd BA, Feig JE, Krishnan P, Sweeny J, Milind M, Moreno P, Mehran R, Kovacic JC, Baber U, Dudley JT, Narula J, Sharma S. Intracoronary Imaging, Cholesterol Efflux, and Transcriptomes After Intensive Statin Treatment: The YELLOW II Study. J Am Coll Cardiol. 2017 Feb 14;69(6):628-640. doi: 10.1016/j.jacc.2016.10.029. Epub 2016 Oct 29. PMID 27989886
- [Background] Johnson KW, Glicksberg BS, Shameer K, Vengrenyuk Y, Krittanawong C, Russak AJ, Sharma SK, Narula JN, Dudley JT, Kini AS. A transcriptomic model to predict increase in fibrous cap thickness in response to high-dose statin treatment: Validation by serial intracoronary OCT imaging. EBioMedicine. 2019 Jun;44:41-49. doi: 10.1016/j.ebiom.2019.05.007. Epub 2019 May 22. PMID 31126891

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 329 Patients were screened with 137 enrolled.
Period: Overall Study
Arm/Group | Treatment
Started | 137
Completed | 110
Not Completed | 27
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 4
Not completed — Death | 2
Not completed — Patient preference | 11
Not completed — Treatment discontinuation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 98
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (19.3)
Hypertension [Count of Participants; unit: Participants] | 127
Previous Percutaneous coronary intervention (PCI) [Count of Participants; unit: Participants] | 97
Previous Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 32
Current smoking [Count of Participants; unit: Participants] | 14
History of smoking [Count of Participants; unit: Participants] | 51
Diabetes [Count of Participants; unit: Participants] | 74
Baseline statin use [Count of Participants; unit: Participants] — High intensity:
  Atorvastin ≥40 mg or Rosuvastatin ≥20 mg
  Moderate intensity:
  Atorvastatin <40 mg or Rosuvastatin <20 mg or Fluvastatin: 40-80 mg or Simvastatin 20-40 mg or Pravastatin 40-80 mg or Lovastatin 40-80 mg or Pitavastatin 1-4 mg
  Low intensity:
  Fluvastatin: 20-40 mg or Simvastatin 10 mg or Pravastatin 10-20 mg or Lovastatin 20 mg Population: 8 statin intolerant patients
  Participants
    number analyzed (Participants) | 129
    High intensity | 91
    Moderate intensity | 38
    Low intensity | 0
Diseased Coronary Vessel Type [Count of Participants; unit: Participants]
  LAD - Left Anterior Descending Artery | 29
  LCX - Left Circumflex Artery | 36
  RCA - Right Coronary Artery | 70
  RI - Ramus Intermedius Artery | 2
Number of diseased vessels [Count of Participants; unit: Participants]
  3 | 4
  2 | 31
  1 | 83
  0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Minimal Fibrous Cap Thickness (FCT)
Description: Changes in the minimal Minimal Fibrous Cap Thickness (FCT) is assessed by Optical Coherence Tomography (OCT) imaging and measured in microns. FCT describes plaque morphology composition.
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Treatment
Number analyzed (Participants) | 110
µm
  Baseline | 70.9 (21.7)
  26 Weeks | 97.7 (31.1)

2. Primary Outcome: Number of Participants With FCT <65 µm
Time Frame: Baseline and 26 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 110
Participants
  Baseline | 53
  26 weeks | 14

3. Primary Outcome: Number of Participants With Increased Fibrous Cap
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 110
Participants | 88

4. Primary Outcome: Change in maxNIRS4mm
Description: Changes in maximal lipid-core burden index within 4 mm (maxLCBI4mm). LCBI4mm is assessed by NIRS and calculated as the fraction of yellow pixels on a chemogram multiplied by 1000. Each pixel on the chemogram represents a probability of lipid presence in the given region; pixels are color-coded on a red-to-yellow color scale, with the low probability of lipid shown as red and the high probability of lipid shown as yellow. Maximal lipid-core burden index is calculated as a fraction of yellow pixels (representing lipid) obtained from the NIRS chemogram multiplied by 1000. It ranges is from 0 to 1000 and represents the amount of lipid in the investigated segment with "0" corresponding to no lipid and "1000" representing all lipid lesion.
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Treatment
Number analyzed (Participants) | 110
index
  Baseline | 306.8 (177.6)
  26 Weeks | 213.1 (168.0)

5. Primary Outcome: Number of Participants With Decreased maxLCBI4mm
Time Frame: 26 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 110
Participants | 86

6. Secondary Outcome: Change in Maximal Lipid Arc
Description: Change in Maximal lipid arc assessed by OCT and measured in degrees.
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Treatment
Number analyzed (Participants) | 110
degrees
  Baseline | 189.1 (73.4)
  26 Weeks | 161.6 (68.7)

7. Secondary Outcome: Change in Lipid Length
Description: Change in Lipid length by OCT, measured in millimeters.
Time Frame: Baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment
Number analyzed (Participants) | 110
mm
  Baseline | 10.4 (6.0)
  26 Weeks | 8.9 (5.6)

8. Secondary Outcome: Change in Lipid Volume Index (LVI)
Description: Change in Lipid Volume Length (LVI) calculated as the average lipid arc multiplied by lipid length assessed by OCT.
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: mm*degrees
Arm/Group | Treatment
Number analyzed (Participants) | 110
mm*degrees
  Baseline | 1259.4 (994.5)
  26 Weeks | 972.0 (855.7)

9. Secondary Outcome: Change in Macrophage Accumulation
Description: Change in the prevalence of Macrophage accumulation (maximum and average) by OCT, a marker of inflammation (expressed as frequency of the presence of macrophages in lesions.)
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Treatment
Number analyzed (Participants) | 110
degrees
  Maximum macrophage arc Baseline | 148.2 (72.5)
  Maximum macrophage arc 26 Weeks | 122.1 (67.7)
  Average macrophage arc Baseline | 83.4 (36.5)
  Average macrophage arc 26 Weeks | 71.2 (32.0)

10. Secondary Outcome: Change in Macrophage Volume Index
Description: Change in the Macrophage Volume Index by OCT, a marker of inflammation (expressed as frequency of the presence of macrophages in lesions.)
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: mm*degrees
Arm/Group | Treatment
Number analyzed (Participants) | 110
mm*degrees
  Baseline | 876.4 (757.6)
  26 Weeks | 590.0 (557.3)

11. Secondary Outcome: Change in Macrophage Length
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment
Number analyzed (Participants) | 110
mm
  Baseline | 9.6 (5.7)
  26 Weeks | 7.6 (5.2)

12. Secondary Outcome: Change in Calcification Accumulation
Description: Change in Calcification accumulation by OCT expressed as frequency of the presence of calcification in lesions.
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Treatment
Number analyzed (Participants) | 110
degrees
  Maximum calcium arc Baseline | 98.6 (55.7)
  Maximum calcium arc 26 Weeks | 98.6 (54.6)
  Average calcium arc Baseline | 61.1 (26.1)
  Average calcium arc 26 Weeks | 61.2 (25.1)

13. Secondary Outcome: Change in Calcium Length
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment
Number analyzed (Participants) | 110
mm
  Baseline | 6.4 (4.9)
  26 Weeks | 6.7 (4.7)

14. Secondary Outcome: Change in Percent Atheroma Volume (PAV)
Description: Change in PAV assessed by Intravascular Ultrasound (IVUS). PAV characterizes coronary plaque burden and calculated as the proportion of total vessel wall volume occupied by atherosclerotic plaque. The percent atheroma volume is calculated as the proportion of total vessel wall volume occupied by atherosclerotic plaque - plaque volume divided by vessel volume and multiplied by 100.
Time Frame: Baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: percent atheroma volume
Arm/Group | Treatment
Number analyzed (Participants) | 110
percent atheroma volume
  Baseline | 51.6 (8.9)
  26 Weeks | 50.2 (8.7)

15. Secondary Outcome: Change in Total Atheroma Volume (TAV)
Description: Change in TAV assessed by IVUS. TAV characterizes the total volume of coronary plaque.
Time Frame: Baseline and 26 Weeks
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Treatment
Number analyzed (Participants) | 110
mm^3
  Baseline | 137.2 (72.8)
  26 Weeks | 131.2 (71.8)

16. Secondary Outcome: Change in PBMC Gene Expression
Description: Change in PBMC gene expression. Messenger RNA sequencing data will be processed using statistical and bioinformatics analyses.
Time Frame: Baseline and 1 year
Reporting Status: Not Posted, anticipated posting 2024-10

ADVERSE EVENTS:
Time Frame: 6 months
Description: Final AE will be reported at 12 months, October 2023 data still being collected
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 2/110
Serious Adverse Events (participants affected / at risk) | 5/110
Other Adverse Events (participants affected / at risk) | 30/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=110)
Myocardial Infarction (Cardiac disorders) | 1
Urgent Revascularization (Cardiac disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=110)
Chest pain/tightness (Cardiac disorders) | 11
Shortness of breath (Cardiac disorders) | 4
Fatigue (Cardiac disorders) | 4
Back/feet pain (Metabolism and nutrition disorders) | 3
Fever (Respiratory, thoracic and mediastinal disorders) | 1
Corneal abrasion (Eye disorders) | 1
Indigestion (Gastrointestinal disorders) | 1
Cold/flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 2
COVID (Respiratory, thoracic and mediastinal disorders) | 1
Groin Pain (Vascular disorders) | 5
Food poisoning (Gastrointestinal disorders) | 1
Nose bleed (Vascular disorders) | 1
Papules (Skin and subcutaneous tissue disorders) | 1
Hives (Skin and subcutaneous tissue disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04710368/Prot_SAP_000.pdf